CLINICAL TRIAL: NCT05804097
Title: Does Increasing Oxygen Nurture Your Symptomatic Ischemic Ulcer Sufficiently?
Acronym: DIONYSIUS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Dirk T. Ubbink, Professor Doctor, Amsterdam UMC, location AMC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL72855.018.20
Record Dates: First submitted 2023-03-24; First posted 2023-04-07 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Vascular Disease; Diabetic Foot Ulcer; Amputation
Keywords: Diabetic Foot Ulcer; Hyperbaric Oxygen; Peripheral Vascular Disease; HBOT; DFU; Major amputation; Diabetes; Ischemia
MeSH Terms: conditions — Peripheral Vascular Diseases; Diabetic Foot; Diabetes Mellitus; Ischemia | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (No Intervention): Control group
- HBOT 20 (Experimental): Patients receiving 20 sessions of concurrent Hyperbaric oxygen treatment
  Interventions: Drug: Hyperbaric oxygen
- HBOT 30 (Experimental): Patients receiving 30 sessions of concurrent Hyperbaric oxygen treatment
  Interventions: Drug: Hyperbaric oxygen
- HBOT 40 (Experimental): Patients receiving at least 40 sessions of concurrent Hyperbaric oxygen treatment
  Interventions: Drug: Hyperbaric oxygen

INTERVENTIONS:
Drug: Hyperbaric oxygen — 90-120 min sessions of hyperbaric oxygen treatment of 2.2-2.5 ATA
  Arms: HBOT 20; HBOT 30; HBOT 40

SUMMARY:
The goal of this multicenter, multi-national, multi-arm, multi-stage, randomized controlled trial, is to determine the added benefit of hyperbaric oxygen treatment (HBOT) in patients with diabetic foot ulcers and peripheral vascular disease. The main question is:

- What is the difference is the major amputation rate between the study arms?

Participants will be randomized to 20, 30 or 40 sessions of HBOT or a control group.

DETAILED DESCRIPTION:
Objective: The primary objective is to assess the (cost-) effectiveness of HBOT in addition to standard wound care and vascular surgical treatment for patients with a DFU and leg ischaemia.

Study design: An international, multi-arm multi-stage (MAMS) design is chosen to conduct an efficient randomised clinical trial. At a planned interim analysis the best performing study arm(s) will be chosen to continue.

Study population: We need up to 544 patients with a Meggitt-Wagner stage 3 or 4 DFU and proven peripheral ischaemia.

Intervention: Patients will be randomised to receive standard care (wound treatment and surgical interventions following international guidelines) with either 0, 20, 30 or at least 40 sessions of HBOT. These sessions will compromise 90-120 minutes of HBOT at a pressure of 2.2-2.5 ATA according to international standards.

Main study parameters/endpoints: The primary endpoint is major amputation rate after 12 months. Secondary objectives are amputation-free survival, wound healing, health-related quality of life and cost-effectiveness of the interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Type I or II diabetes
2. One or more deep and clinically infected lower extremity ulcers, classified as Meggitt-Wagner class 3 or 4, Texas class 2C, 3C, 2D or 3D, or WIfI class W>1, I>1 and fI>0), present for at least 4 weeks or after a minor amputation because of a previously existing ischaemic DFU on a toe or forefoot. In case more than one ulcer is present, the largest will be observed as target ulcer
3. Leg ischaemia, characterized by a highest ankle systolic blood pressure < 70 mmHg, or a toe systolic pressure < 50 mmHg or a TcpO2 < 40 mmHg
4. Complete assessment of peripheral arterial lesions from the aorta to the pedal arteries with duplex ultrasonography, magnetic resonance angiography, computed tomography angiography and/or intraarterial digital subtraction angiography of the ipsilateral leg
5. Patients have to be discussed in, and included after a multidisciplinary consultation.
6. Adults
7. Written informed consent

Exclusion Criteria:

1. Chronic Obstructive Pulmonary Disease (COPD) GOLD IV
2. Treatment with chemotherapy, immunosuppressive drugs or systemic corticosteroids within last 3 months, as this interferes with normal wound healing
3. End-stage renal disease requiring dialysis
4. Metastasized malignancy
5. Left ventricular failure with ejection fraction (EF) <20% or external pacemaker
6. Recent thoracic surgery or middle ear surgery
7. Severe epilepsy
8. Uncontrollable high fever
9. Pregnancy
10. Insufficient proficiency of local language/English, or inability to complete the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Major Amputations | 12 months after inclusion
  Major amputations, defined as below the knee or above the knee amputations

SECONDARY OUTCOMES:
Amputation-free survival | Complete follow-up (up to 3 years)
  Time without amputation
Health-related quality of life | Complete follow-up (up to 3 years)
  Quality of life based on various questionnaires (objective)
Complete wound healing | 12 months after inclusion
  Complete wound healing
Pain scores | 12 months after inclusion
  Pain scores taken by VAS questionnaire
Need for additional (vascular) interventions | Complete follow-up (up to 3 years)
  Vascular interventions performed during time of inclusion
Cost-effectiveness and budget impact | Complete follow-up (up to 3 years)
  Costs of healthcare resources, including HBOT, related to the total number of eligible patients for HBOT per year.
  QALYs, based on EQ-5D-5L
Mortality | Complete follow-up (up to 3 years)
  Mortality
Patients perception of improvement | Complete follow-up (up to 3 years)
  Quality of life based on various questionnaires (subjective)
TcpO2 before, during and after HBOT | During intervention period
  Measurements of TcpO2 surrounding HBOT treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, Noord-Hollad, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after deidentification (text, tables, figures and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication and 10 years following article publication.
Access Criteria: Researchers who provide a scientifically good reason to require access. If approved data can be shared after the signing a Data Access Agreement.

REFERENCES:
- [Derived] Brouwer R, van der Peet R, Hoencamp R, Koelemay M, van Dieren S, van Hulst R, Ubbink D. DIONYSIUS trial: "Does increasing oxygen nurture your symptomatic ischaemic ulcer sufficiently?" Study protocol for an international multicentre randomised trial. BMJ Open. 2023 May 25;13(5):e063503. doi: 10.1136/bmjopen-2022-063503. PMID 37230523